CLINICAL TRIAL: NCT07042139
Title: A Randomized Controlled Trial Comparing No Reduction to Closed Reduction for Distal Radius Fractures in Patients 65 Years and Older (DISCLOSE Trial): A Study Protocol
Brief Title: No Reduction Compared to Closed Reduction for Distal Radius Fractures in Patients Over 65 or Older
Acronym: DISCLOSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Kuopio University Hospital (Other); Viborg Regional Hospital (Other); Karolinska University Hospital (Other); Helsinki University Central Hospital (Other); Tartu University Hospital (Other); Pori Central Hospital (Unknown); Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R25001
Record Dates: First submitted 2025-04-14; First posted 2025-06-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Distal Radius Fracture; Casting; Closed Reduction
Keywords: distal radius fracture; casting; closed reduction; nonoperative treatment; DISCLOSE trial
MeSH Terms: conditions — Wrist Fractures | interventions — Closed Fracture Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: To minimize the risk of biased interpretation, the trial results will be analyzed using a blinded data interpretation process, in which the statistician will remain masked to the group allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed Reduction (Active Comparator): Closed reduction and casting after distal radius fracture
  Interventions: Procedure: Closed Reduction; Other: Casting
- No Reduction (Experimental): Casting without reduction after distal radius fracture
  Interventions: Procedure: No reduction; Other: Casting

INTERVENTIONS:
Procedure: No reduction — No reduction
  Arms: No Reduction
Procedure: Closed Reduction — Closed reduction
  Arms: Closed Reduction
Other: Casting — Dorsal cast

SUMMARY:
DISCLOSE trial is a randomized controlled trial including 532 participants with low-energy distal radius fractures. The primary objective is to evaluate whether casting without prior closed reduction is equivalent to casting following closed reduction with respect to wrist-related pain and disability, as measured by the Patient-Rated Wrist Evaluation (PRWE) score at 12 months, in patients aged 65 years or older with a displaced distal radius fracture.

* Primary endpoint will be PRWE at 12 months
* Follow-up visits are scheduled at 3 and 12 months. 5-year follow-up will be considered as an exploratory endpoint

DETAILED DESCRIPTION:
Interventions:

No reduction: In the no reduction group, a dorsal cast is applied to the patient's wrist after the initial radiograph. Following casting, a control radiograph will be taken. Active range of motion exercises for the fingers and light use of the hand are recommended immediately.

Closed reduction: Distal radius fracture reduction is performed in the emergency department under local anaesthetic, with lidocaine infiltrated into the fracture site. Closed reduction is performed by the on-call physician who is responsible for the patient's treatment. Post-reduction radiographs are then taken to assess fracture alignment, although the findings do not influence the treatment of the patient. The follow-up visits, cast removal, and exercise protocol are identical to those inof the no reduction group.

In both groups, the cast will be removed after 5 weeks at either the health center or the hospital's outpatient clinic, in accordance with the local treatment protocol. Following cast removal, patients will be advised to resume everyday use of the injured wrist without restrictions. No radiographs will be taken during the casting period or before the 3-month follow-up.

Observational arm (not part of the randomised equivalence trial): Eligible patients who decline participation in the randomisation will be offered the opportunity to join an observational group. The patients will receive standard care (closed reduction and casting) and will provide consent for follow-up. Reduction of the DRF is performed in the emergency department and post-reduction radiographs will be taken. The observational groups will be treated according to local treatment protocols. Patients in the observational cohort will be followed at the same time points using the same outcome measures as the randomised group. Study follow-up of the observational group will be organized remotely.

Blinding: Recruiting will start at July 2025.Due to the nature of the intervention, the participants will not be blinded. Recruiting personnel will only have access to the randomisation module within the electronic REDCap (Research Electronic Data Capture, https://www.project-redcap.org/) software. The outcome assessors (study nurse or orthopaedic resident or specialist) who collect the baseline data and outcome measures from the follow-up visits will be blinded to the randomisation result. Furthermore, the study personnel involved in the follow-up visits will remain blinded to the randomisation results, as the results will be hidden in REDCap.

Follow-up: Participants will meet a research personnel or coordinator study nurse at the 3-month and 12-month time points. At the 3-month time point, radiographs will be taken. Thereafter, no additional radiographic follow-ups will be organized. Follow-up appointments will be carried out according to the preferences of the participants. For example, all patients will be invited to attend an in-person follow-up visit; however, if this is unsuitable, the follow-up will be conducted remotely via telephone or email link by a blinded study nurse. In the remote option, the accelerometer wristbands will be sent to the participants by regular mail. By offering a remote option, we aim to minimise the number of participants unavailable for follow-up. The participants will receive follow-up questionnaires via email or regular mail prior to their follow-up appointment. If they decline to complete the questionnaires, outcomes will be collected via a telephone interview. The research data will be saved in a database using the online patient management program REDCap. The 5-year follow-up will be conducted by phone.

Rehabilitation: All patients presenting with unsettling symptoms will undergo physiotherapy rehabilitation for up to one year, as in standard care. If the symptoms do not improve during this period, the patient will be referred to an orthopaedic surgeon or hand surgeon for further evaluation where necessary procedures, such as a computed tomography (CT) scan and, in some cases corrective osteotomy, will be considered.

Sample size and power considerations: The sample size was determined based on an equivalence design with an equal allocation ratio (1:1). Based on the MID for PRWE of 11.5 points, the equivalence margin was set at 6 points. This represents the maximum acceptable difference in means between the groups to still be able to consider the groups as equivalent. Based on the findings of previous studies, the standard deviation of the outcome (PRWE) variable was estimated to be 21.9. Using these parameter estimates, a total sample size of 532 participants (266 per group) will provide 90% power to demonstrate equivalence between groups on the primary endpoint, assuming a true mean difference of < 0.01, a common standard deviation of 21, and equivalence margins of -6 to 6 on the PRWE score. The calculation was based on a 2-sided 90% confidence interval (α = 0.05) and used the exact method for two-sample means under normal distribution assumptions.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Independent living patients
* Displaced distal radius fracture (AO/OTA 23A/23C) with 15-40 degree dorsal angulation, and/or of shortening of the radius for more than 2 mm.
* Associated ulnar styloid fracture is permitted
* Low energy injury, (fall from <1 m)

Exclusion Criteria:

* Patient unable to provide consent
* Patients who are actively working in a paid position
* Volar angulation, partial articular fractures (AO/OTA 23B)
* Concomitant fracture of the ulna proximal to the base of the styloid process
* Associated fracture or dislocation in any other body part that would affect the use of the injured distal radius
* Distal radius fractures in both arms
* Open injury, Gustilo 2 or higher
* No bony contact between the main fragments
* High energy injuries

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2033-07-01 (Estimated)

PRIMARY OUTCOMES:
PRWE | 12 months
  Primary outcome will be the Patient Rated Wrist Evaluation (PRWE) at 12 months. PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. The questionnaire consists of two subscales (pain and function), and the score ranges from 0 (no disability) to 100 (severe disability).

SECONDARY OUTCOMES:
Pain (NRS) | 3 months and 12 months
  The Numeric Rating Scale (NRS) is a subjective measure of acute pain. The Numeric Rating Scale (NRS) for Pain is a validated 11-point numerical rating scale for acute and chronic pain with terminal descriptors of 0 (no pain) and 10 (worst pain possible). Patients will be asked to evaluate their perceived pain during the previous 7 days.
PASS | 3 months and 12 months
  Patient satisfaction will be measured using the patient-acceptable symptom state (PASS). The questionnaire includes the following question: Considering all the different ways your injury is affecting you, if you would remain in this state, do you feel that your current state is satisfactory (Yes/No)?
EQ-5D-5L- Quality of life | 3 months and 12 months
  EuroQol 5-dimension 5-level health-related quality of life questionnaire (EQ-5D-5L). It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. We will use the EQ-5D-5L Index score, which is calculated based on each dimension using population-specific preference weights and will be reported on a scale from less than 0 to 1.
Serious adverse events | 3 months and 1 year
  Serious adverse events include, but are not limited to: late surgical interventions such as corrective osteotomy or internal fixation due to symptomatic nonunion; tendon repair; carpal tunnel release; acute nerve injury confirmed by electroneuromyography; and any other adverse event that results in hospitalisation, prolongation of existing hospitalisation, is life-threatening, or leads to persistent or significant disability (for example CRPS) or incapacity. Serious adverse events will be assessed at 3- and 12-months timepoints.
Cosmesis | 3 months
  Participants are asked to complete questionnaire about wrist cosmesis. Does the appearance of the wrist bother you? (yes/no)

OTHER OUTCOMES:
Radiographic measurements | Baseline and 3 months
  Radiographic parameters will be collected from radiographs taken at baseline and after casting. Control radiographs will be taken at the 3-month time point where the loss of reduction is measured. Radiographic measurements will include dorsal angulation (degrees), ulnar variance (mm), radial inclination (degrees), step-off in the articular surface (mm), and intra-articular gap (mm)
Tri-Axial Accelerometry (Published separately) | 3 and 12 months
  The upper-limb physical activity of the participants will be measured using a tri-axial (Axivity Ltd, Newcastle upon Tyne, UK) accelerometer. Activity is divided into 4 activity levels (inactive, light, moderate and vigorous), and also sleeping time is counted and recorded.
Cost-effectiveness (Published separately) | 12 months
  Included unit cost components include hospital stays and outpatient visits, including imaging, surgical and anesthetic procedures, physiotherapy, complication management and re-operations and cast changes. Costs will be obtained directly from patients through questionnaires administered at the 3 and 12 month follow-up, and from medical records. Cost data will be derived from the NordDRG classification system. Using the mean costs and mean health outcomes for each cohort, the incremental cost per quality-adjusted life-year (QALY) gained will be calculated.
5 year exploratory endpoint (Published separately) | 5-year
  PRWE, pain (NRS), quality of life, patient satisfaction (PASS), serious adverse events, and mortality will be assessed at 5 years and are exploratory endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kärnä, MD, Principal Investigator — Tampere University Hospital; Ville Ponkilainen, Principal Investigator — Tampere University Hospital; Antti Launonen, Principal Investigator — Tampere University Hospital
Locations (10):
- Viborg regional Hospital, Viborg, Denmark
- Tartu University Hospital, Tartu, Estonia
- Finland (7):
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Helsinki University Hospital, Helsinki, Uusimaa
  - Kanta-Häme Central Hospital, Hämeenlinna
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Pori Central Hospital, Pori
  - Turku University Hospital, Turku
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to restrictions under Finnish data protection regulations, which limit the sharing of sensitive personal data, even in de-identified form, without specific consent or legal basis.

REFERENCES:
- [Derived] Karna L, Ponkilainen V, Reito A, Ostergaard H, Brorson S, Tootsi K, Paasikallio K, Senholt T, Li Y, Heikkinen J, Kukkonen J, Ryhanen J, Christensen R, Mattila VM, Launonen AP. Effect of no reduction versus closed reduction on distal radius fractures in adults aged 65 years and older: a protocol for the DISCLOSE randomised equivalence trial. BMJ Open. 2025 Oct 16;15(10):e108511. doi: 10.1136/bmjopen-2025-108511. PMID 41101953

DOCUMENTS (1):
  • Study Protocol (2025-07-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT07042139/Prot_000.pdf